CLINICAL TRIAL: NCT02344004
Title: A Randomized, Open-label, Multicenter Study of Liposomal Amikacin for Inhalation (LAI) in Adult Patients With Nontuberculous Mycobacterial (NTM) Lung Infection Caused by Mycobacterium Avium Complex (MAC) That Are Refractory to Treatment
Brief Title: Study to Evaluate Efficacy of LAI When Added to Multi-drug Regimen Compared to Multi-drug Regimen Alone
Acronym: CONVERT
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Insmed Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: INS-212; 2014-005010-31 (EudraCT Number)
Record Dates: First submitted 2015-01-09; First posted 2015-01-22 (Estimated); Results first posted 2018-11-20 (Actual); Last update posted 2020-05-07 (Actual); Status verified 2020-02

CONDITIONS: Mycobacterium Infections, Nontuberculous
Keywords: ALIS; ARIKAYCE
MeSH Terms: conditions — Mycobacterium Infections, Nontuberculous | interventions — Inhalation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Multi-drug Regimen (No Intervention): Participants received their already prescribed anti-mycobacterial regimen (based on the 2007 American Thoracic Society/Infectious Diseases Society of America [ATS/IDSA] Guidelines)
- LAI + Multi-drug Regimen (Experimental): Participants received LAI 590 mg QD in addition to their already prescribed anti-mycobacterial regimen (based on the 2007 ATS/IDSA Guidelines)
  LAI 590 mg QD, administered by inhaling drug product that had been aerosolized in an eFlow nebulizer over approximately 14 minutes
  Interventions: Drug: LAI (Liposomal Amikacin for Inhalation) 590 mg

INTERVENTIONS:
Drug: LAI (Liposomal Amikacin for Inhalation) 590 mg — LAI 590 mg QD, administered by inhaling drug product that had been aerosolized in an eFlow nebulizer over approximately 14 minutes.
  Other Names: ALIS (Amikacin Liposome Inhalation Suspension); ARIKAYCE®
  Arms: LAI + Multi-drug Regimen

SUMMARY:
A study to evaluate the effectiveness of Liposomal Amikacin for Inhalation (LAI) 590 mg administered once daily (QD) when added to multi-drug regimen (MDR) in participants with Nontuberculous Mycobacterial (NTM) lung infection caused by Mycobacterium Avium Complex (MAC) that were refractory to treatment.

Participants were randomized 2:1 to LAI 590 mg administered QD + MDR or MDR alone.

DETAILED DESCRIPTION:
This is a randomized, open-label, multicenter study of LAI in adult participants with NTM lung infections caused by MAC that were refractory to treatment. Participants received either LAI 590 mg administered QD by inhalation plus a multidrug regimen, hereafter referred to as LAI + MDR or a multidrug regimen alone, hereafter referred to as MDR alone for a minimum of 8 months. Participants who demonstrated culture conversion by Month 6 went on to complete a treatment course of 12 months, starting from the first of 3 negative cultures that defined culture conversion.

Sputum culture results were made available to the site after the Month 6 sputum result was known, in time for the Month 8 visit. Prior to the Month 8 visit, the culture results from Baseline to Month 6 inclusively were blinded to the site and Sponsor. The results were blinded to reduce the potential for bias in an open-label study. At Month 8 (-28 to +7 days), after all sputum culture results were made available to the site only, up to and including Month 6, participants were assessed as converters or non-converters.

A converter was defined as a participant who had 3 consecutive monthly MAC-negative sputum cultures at any time within the first 6 months of the study.

"Relapse or recurrence" was defined as having MAC-positive sputum cultures in liquid broth media (agar negative) for 3 or more consecutive months, or having at least 1 MAC-positive sputum culture on solid media (agar positive) after achieving culture conversion.

A non-converter was defined as a participant who did not have 3 consecutive monthly MAC-negative sputum cultures at any time within the first 6 months of the study.

All converters remained in the study. Converters who, after culture conversion, subsequently had MAC-positive sputum cultures in liquid broth media (agar negative) for 1 or 2 consecutive months only by Month 6 also remained in the study. Participants who remained in the study continued their randomized treatment regimen until they completed a total of 12 months of treatment (EOT), starting from the first of 3 negative cultures that defined culture conversion. These participants returned after the EOT visit for 28 days, 3, 6, and 12 months off-treatment follow-up visits. The 12 months off-treatment follow-up visit was the end of study (EOS) visit. No NTM treatment was administered during the off-treatment phase.

At Month 8, all non-converters as assessed at the Month 6 visit were discontinued from Study INS-212. Participants who experienced a relapse or recurrence by Month 6 also discontinued from Study INS-212 at their Month 8 visit. These participants were potentially eligible to enter a separate open-label study of LAI (Study INS-312), provided all entry criteria were met for that study.

ELIGIBILITY:
Inclusion Criteria:

1. Be continually positive for MAC on sputum culture while adhering to a multi-drug treatment regimen for a minimum duration of 6 months which is either ongoing or was completed no more than 12 months before screening
2. Be diagnosed with MAC NTM lung infection with evidence of nodular bronchiectasis and/or fibrocavitary disease by chest CT
3. Be willing to adhere to multi-drug treatment regimen during the course of the study

Exclusion Criteria:

1. Patients with cystic fibrosis
2. Positive pregnancy test or lactation at screening. All women of child bearing potential will be tested. Women not of childbearing potential are defined as postmenopausal (i.e., amenorrheic for at least 1 year), or surgically or naturally sterile.
3. Active pulmonary tuberculosis requiring treatment at screening
4. History of lung transplantation
5. Prior exposure to LAI (including clinical study).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 336 (Actual)
Dates: Start 2015-05-27 (Actual); Primary Completion 2018-07-03 (Actual); Study Completion 2019-04-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gina Eagle, MD, Study Director — Insmed Incorporated

REFERENCES:
- [Derived] Yamazaki Y, Nakagawa T, Jumadilova Z, Yuen D, Villa R, Hasegawa N. Management and Resolution of Hypersensitivity Pneumonitis-Related Events in Japanese Patients Treated with Amikacin Liposome Inhalation Suspension in the CONVERT and INS-312 Clinical Trials. Infect Dis Ther. 2025 Nov 4. doi: 10.1007/s40121-025-01247-7. Online ahead of print. PMID 41186908
- [Derived] Morimoto K, Nonaka M, Yamazaki Y, Nakagawa T, Takasaki J, Tsuyuguchi K, Kitada S, Jumadilova Z, Yuen DW, Ciesielska M, Hasegawa N. Amikacin liposome inhalation suspension for Mycobacterium avium complex pulmonary disease: A subgroup analysis of Japanese patients in the randomized, phase 3, CONVERT study. Respir Investig. 2024 Mar;62(2):284-290. doi: 10.1016/j.resinv.2023.12.012. Epub 2024 Jan 25. PMID 38277865
- [Derived] Griffith DE, Thomson R, Flume PA, Aksamit TR, Field SK, Addrizzo-Harris DJ, Morimoto K, Hoefsloot W, Mange KC, Yuen DW, Ciesielska M, Wallace RJ Jr, van Ingen J, Brown-Elliott BA, Coulter C, Winthrop KL; CONVERT Study Group. Amikacin Liposome Inhalation Suspension for Refractory Mycobacterium avium Complex Lung Disease: Sustainability and Durability of Culture Conversion and Safety of Long-term Exposure. Chest. 2021 Sep;160(3):831-842. doi: 10.1016/j.chest.2021.03.070. Epub 2021 Apr 19. PMID 33887244
- [Derived] Rubino CM, Onufrak NJ, van Ingen J, Griffith DE, Bhavnani SM, Yuen DW, Mange KC, Winthrop KL. Population Pharmacokinetic Evaluation of Amikacin Liposome Inhalation Suspension in Patients with Treatment-Refractory Nontuberculous Mycobacterial Lung Disease. Eur J Drug Metab Pharmacokinet. 2021 Mar;46(2):277-287. doi: 10.1007/s13318-020-00669-7. Epub 2021 Feb 17. PMID 33595792
- [Derived] Griffith DE, Eagle G, Thomson R, Aksamit TR, Hasegawa N, Morimoto K, Addrizzo-Harris DJ, O'Donnell AE, Marras TK, Flume PA, Loebinger MR, Morgan L, Codecasa LR, Hill AT, Ruoss SJ, Yim JJ, Ringshausen FC, Field SK, Philley JV, Wallace RJ Jr, van Ingen J, Coulter C, Nezamis J, Winthrop KL; CONVERT Study Group. Amikacin Liposome Inhalation Suspension for Treatment-Refractory Lung Disease Caused by Mycobacterium avium Complex (CONVERT). A Prospective, Open-Label, Randomized Study. Am J Respir Crit Care Med. 2018 Dec 15;198(12):1559-1569. doi: 10.1164/rccm.201807-1318OC. PMID 30216086

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at 127 sites in 18 countries.
Pre-assignment Details: Participant flow table reflects the disposition through end of the study (Month 28).
  The deaths under Reasons for Discontinuation reflect the primary reason (according to investigator's judgment) that the participant discontinued and does not represent all deaths in the trial.
Groups:
- LAI + Multi-drug Regimen: Participants received Liposomal Amikacin for Inhalation (LAI) 590 mg once daily (QD) in addition to their already prescribed anti-mycobacterial regimen (based on the 2007 American Thoracic Society/Infectious Diseases Society of America [ATS/IDSA] Guidelines); LAI 590 mg QD, administered by inhaling drug product that had been aerosolized in an eFlow nebulizer over approximately 14 minutes
- Multi-drug Regimen: Participants received their already prescribed anti-mycobacterial regimen (based on the 2007 ATS/IDSA Guidelines)
Period: Overall Study
Arm/Group | LAI + Multi-drug Regimen | Multi-drug Regimen
Started | 224 | 112
Completed | 163 | 98
Not Completed | 61 | 14
Not completed — Adverse Event | 11 | 1
Not completed — Death | 9 | 7
Not completed — Physician Decision | 4 | 1
Not completed — Withdrawal by Subject | 22 | 5
Not completed — Rescue Medication | 2 | 0
Not completed — Other Not Specified | 12 | 0
Not completed — Protocol Violation | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- LAI + Multi-drug Regimen: Participants received LAI 590 mg QD in addition to their already prescribed anti-mycobacterial regimen (based on the 2007 ATS/IDSA Guidelines); LAI 590 mg QD, administered by inhaling drug product that had been aerosolized in an eFlow nebulizer over approximately 14 minutes
- Total: Total of all reporting groups
Arm/Group | LAI + Multi-drug Regimen | Multi-drug Regimen | Total
Number analyzed (Participants) | 224 | 112 | 336
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.6 (9.59) | 64.9 (10.16) | 64.7 (9.77)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 165 | 68 | 233
  Male | 59 | 44 | 103
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 10 | 5 | 15
  Not Hispanic or Latino | 211 | 102 | 313
  Unknown or Not Reported | 3 | 5 | 8
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 58 | 25 | 83
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Black or African American | 3 | 3 | 6
  White | 158 | 77 | 235
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 3 | 6 | 9
If female, is participant of childbearing potential? [Count of Participants; unit: Participants] — Population: 165/224 female participants in the LAI + Multi-drug regimen arm
  68/112 female participants in the Multi-drug regimen arm
  Participants
    number analyzed (Participants) | 165 | 68 | 233
    Yes | 13 | 6 | 19
    No | 152 | 62 | 214
If not childbearing potential, specify [Count of Participants; unit: Participants] — Population: 152/224 female participants not of childbearing potential in the LAI + Multi-drug regimen arm
  62/112 female participants not of childbearing potential in the Multi-drug regimen arm
  Participants
    number analyzed (Participants) | 152 | 62 | 214
    Postmenopausal | 114 | 50 | 164
    Surgically Sterile | 38 | 12 | 50
    Naturally Sterile | 0 | 0 | 0
Region [Count of Participants; unit: Participants]
  North America | 104 | 55 | 159
  Asia (excluding Japan) | 14 | 6 | 20
  Japan | 34 | 14 | 48
  Rest of World | 72 | 37 | 109
Multidrug regimen prior to enrollment [Count of Participants; unit: Participants]
  On treatment | 201 | 101 | 302
  Off treatment for at least 3 months | 23 | 11 | 34
Smoking status (includes e-cigarettes) [Count of Participants; unit: Participants]
  Current smoker | 26 | 10 | 36
  Not a current smoker | 198 | 102 | 300
Prior nebulized IV amikacin [Count of Participants; unit: Participants] — Participants who had received prior nebulized IV amikacin
  Participants | 24 | 15 | 39

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Achieving Culture Conversion by Month 6 in the Liposomal Amikacin for Inhalation (LAI) + Multi-drug Regimen (MDR) Arm Compared to the MDR Alone Arm
Description: Sputum specimens were collected at Screening (Visit 1), Baseline (Visit 2), and at Visits 3 (Month 1) through 8 (Month 6). A negative culture result reflected a negative culture result for all sputum samples collected at each visit. Participants met the primary endpoint of culture conversion by Month 6 if they had 3 consecutive monthly MAC-negative sputum cultures during the first 6 months of the study. A participant needed to achieve the first of 3 consecutive negative sputum cultures (that defined culture conversion) by Month 4 in order to meet the primary endpoint by Month 6. Each participant in the intent to treat (ITT) population (ie, all randomized participants) was classified as either a converter or non-converter by Month 6.
Time Frame: by Month 6
Population: The ITT population was the set of all randomized participants. Participants were classified according to their assigned treatment. There was a total of 336 participants in the ITT population, including 224 participants in the LAI + MDR arm and 112 participants in the MDR alone arm.
Measure: Count of Participants; unit: Participants
Groups:
- LAI + Multi-drug Regimen: Participants received LAI 590 mg once daily (QD) in addition to their already prescribed anti-mycobacterial regimen (based on the 2007 ATS/IDSA Guidelines); LAI 590 mg QD, administered by inhaling drug product that had been aerosolized in an eFlow nebulizer over approximately 14 minutes
Arm/Group | LAI + Multi-drug Regimen | Multi-drug Regimen
Number analyzed (Participants) | 224 | 112
Participants
  Converter | 65 | 10
  Non-Converter | 159 | 102
Statistical Analysis 1: Comparison: LAI + Multi-drug Regimen vs Multi-drug Regimen; The proportion of participants achieving culture conversion by Month 6 was analyzed using the Cochran-Mantel-Haenszel test, stratified by smoking status and prior multi-drug regimen. The treatment comparison was tested at two-sided significance level of 0.05. The null hypothesis assumed that culture conversion by Month 6 is independent of treatment, and the alternative hypothesis assumed that culture conversion by Month 6 is associated with treatment; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel; The final analysis of the primary endpoint, the number of participants achieving culture conversion at by Month 6, was performed after the last participants completed Month 6 and his/her Month 6 sputum culture result was available

2. Primary Outcome: Number of Participants Achieving Durable Culture Conversion Through 3 Months Off Treatment in the LAI + MDR Arm Compared to the MDR Arm Alone
Description: Sputum specimens were collected at screening, baseline (Day 1), during treatment, and at Months 1, 3, 6, and 12 months off treatment. Culture conversion with durability was defined as achieving culture conversion by Month 6 and then having no more than 2 consecutive broth positive cultures and no Agar positive culture up to 3 months off treatment. Converters with missing broth or Agar sputum culture result after Month 6 up to 3 months off treatment were considered as not achieving culture conversion with durability except those participants who are unable to produce sputum despite reasonable efforts, as reported by source documentation. Participants who had relapse/recurrence, had "rescue" medication and/or died before reaching 3 months off treatment were considered as not achieving culture conversion with durability.
Time Frame: up to Month 19
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | LAI + Multi-drug Regimen | Multi-drug Regimen
Number analyzed (Participants) | 224 | 112
Participants
  Durable Conversion | 36 | 0
  Non-Durable Conversion | 188 | 112
Statistical Analysis 1: Comparison: LAI + Multi-drug Regimen vs Multi-drug Regimen; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel

3. Secondary Outcome: Change From Baseline (Day 1) to Month 6 in the Six-Minute Walk Test (6MWT) Distance in the LAI + MDR Arm Compared to the MDR Alone Arm
Description: A 6-minute walk assessment of exertional capability was performed at Baseline (Day 1) and at Month 6. The standardized protocol based on the ATS guidelines was used. The 6MWT was conducted by a site member who was blinded to the participant's open-label treatment assignment. The analysis of the change from Baseline (Day 1) to Month 6 in the 6MWT distance was performed after the last participant completed Month 6 and his/her 6MWT distance data were available.
Time Frame: at Month 6
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: meters
Arm/Group | LAI + Multi-drug Regimen | Multi-drug Regimen
Number analyzed (Participants) | 224 | 112
meters
  Baseline: number analyzed (Participants) | 223 | 112
  Baseline | 424.2 (1.12) | 420.9 (0.48)
  Month 6: number analyzed (Participants) | 223 | 112
  Month 6 | 420.6 (4.73) | 420.3 (2.57)
  Change from Baseline to Month 6: number analyzed (Participants) | 223 | 112
  Change from Baseline to Month 6 | -3.6 (3.25) | -0.5 (4.20)
Statistical Analysis 1: Comparison: LAI + Multi-drug Regimen vs Multi-drug Regimen; This was analyzed using a mixed model repeated measures (MMRM) analysis of change from Baseline at Months 4&6. MMRM included treatment, month, treatment-by-month interaction, combination of smoking status & prior MDR (4 levels: Yes/Yes, Yes/No, No/Yes, and No/No) as fixed factors, baseline 6MWD as a covariate & baseline 6MWD-by-month interaction. An unstructured covariance matrix was used for the MMRM; Test type: Superiority; p = 0.7804, Mixed Model Repeated Measures (MMRM); * Baseline is defined as the last non-missing value prior to first dose of study drug. * Statistics were obtained from an mixed-effects model repeated measures (MMRM) model with pattern-mixture modeling of missing values due to dropout, which included treatment, month, the treatment-by-month interaction, and the combination of smoking status and prior multidrug regimen as fixed factors, the baseline 6MWT distance as a covariate and baseline 6MWT distance-by-month interaction. MMRM included postbaseline data through Month 6. * For baseline, n is the number of participants with a baseline score and at least 1 postbaseline score. For Month 6, n is the number of participants with a baseline score and a postbaseline score at the summarized visit

4. Secondary Outcome: Time to Culture Conversion by Month 6 in the LAI + MDR Arm Compared to the MDR Alone Arm
Description: The time to culture conversion was defined by the date of the first of at least 3 consecutive monthly culture specimens that were Mycobacterium avium complex (MAC)-negative.
  The 25th percentile time to conversion is the estimated time taken for 25% of participants to convert.
  The 50th percentile time to conversion is the estimated time taken for 50% of participants to convert.
Time Frame: by Month 6
Population: There was a total of 336 participants in the ITT population, including 224 participants in the LAI + MDR arm and 112 participants in the MDR alone arm.
Measure: Number (95% Confidence Interval); unit: months
Arm/Group | LAI + Multi-drug Regimen | Multi-drug Regimen
Number analyzed (Participants) | 224 | 112
months
  25th Percentile | 2.13 [1.83 to 3.87] | NA [NA to NA] — The 25th percentile time to conversion could not be estimated due to an insufficient proportion of patients achieving culture conversion by Month 6.
  50th Percentile | NA [NA to NA] — The 50th percentile time to conversion could not be estimated due to an insufficient proportion of patients achieving culture conversion by Month 6. | NA [NA to NA] — The 50th percentile time to conversion could not be estimated due to an insufficient proportion of patients achieving culture conversion by Month 6.
Statistical Analysis 1: Comparison: LAI + Multi-drug Regimen vs Multi-drug Regimen; Kaplan Meier estimates for the distribution of time to culture conversion were constructed for treatment arms. The treatment comparison was made using the stratified log rank test for the ITT population. The estimated median time to culture conversion for each treatment arm was not estimable. The time to culture conversion was analyzed using Cox regression model to estimate hazards ratio; Test type: Superiority; p < 0.0001, Regression, Cox; Cox Proportional Hazard = 3.92, 95% CI 2-sided [2.01 to 7.63]

5. Secondary Outcome: Number of Participants Achieving Sustained Culture Conversion at the End of Treatment (EOT) in the LAI + MDR Arm Compared to the MDR Arm Alone
Description: Sustained conversion was evaluated in participants who completed at least 12 months of treatment from the start of culture conversion. Sustained conversion was defined as conversion (3 consecutive negative monthly sputum samples) by Month 6 with no positive agar media culture or no more than 2 broth media cultures up to and including the time point. Participants who did not convert were considered non-sustained conversions.
Time Frame: up to Month 16
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | LAI + Multi-drug Regimen | Multi-drug Regimen
Number analyzed (Participants) | 224 | 112
Participants
  Sustained Conversion | 41 | 3
  Non-Sustained Conversion | 183 | 109

6. Secondary Outcome: Change in 6-Minute Walk Test (6MWT) Distance at EOT in the LAI Arm Compared to a Multi-drug Regimen Alone
Description: A 6-minute walk assessment of exertional capability was performed at Baseline (Day 1) and up to EOT or Month 16. The standardized protocol based on the ATS guidelines was used. The 6MWT was conducted by a site member who was blinded to the participant's open-label treatment assignment.
Time Frame: up to Month 16
Population: Due to the widely varying timepoints that makeup the EOT visit, this was not considered an appropriate analysis and was not performed.
Arm/Group | LAI + Multi-drug Regimen | Multi-drug Regimen
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: Change From Baseline (Day 1) at Month 6 in the St. George's Respiratory Questionnaire (SGRQ) Total Score
Description: The SGRQ was completed before administration of study drug at Baseline (Day 1) and Months 3, 6, 8, and 12, and at the EOT visit and the 3 months off treatment visit. The SGRQ is a self-administered questionnaire that has been validated in participants with airways disease, specifically in participants with bronchiectasis. The SGRQ assesses health-related quality of life in participants with chronic pulmonary disease by evaluating 3 health domains: symptoms (distress caused by respiratory symptoms); activity (effects of disturbances on mobility and physical activity); and impacts (the effect of disease on factors such as employment, personal control of one's health, and need for medication). A composite total score is derived as the sum of domain scores for symptoms, activity, and impact (0 = best possible score and 100 = worst possible score). A within patient reduction from baseline in score of 4 units is generally recognized as a clinically meaningful improvement in quality of life.
Time Frame: at Month 6
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | LAI + Multi-drug Regimen | Multi-drug Regimen
Number analyzed (Participants) | 224 | 112
score on a scale
  SGRQ Total Score at Baseline:: number analyzed (Participants) | 168 | 104
  SGRQ Total Score at Baseline: | 36.555 (21.3777) | 38.409 (21.5753)
  SGRQ Total Score at Month 6:: number analyzed (Participants) | 169 | 106
  SGRQ Total Score at Month 6: | 38.715 (22.3559) | 37.368 (23.6868)
  Change from Baseline to Month 6:: number analyzed (Participants) | 168 | 104
  Change from Baseline to Month 6: | 2.009 (13.4128) | -1.312 (11.6216)

ADVERSE EVENTS:
Time Frame: Treatment-emergent adverse events (AEs) were assessed at Baseline (Day 1) and all subsequent study visits through Month 28 (end of study).
Description: The analysis population consisted of the safety population, defined as all participants who received at least 1 dose of either LAI+ MDR (multi-drug regimen) or MDR alone.
  Participants counted in all-cause mortality constitutes all deaths, regardless of whether or not there was an adverse event.
Arm/Group | LAI + Multi-drug Regimen | Multi-drug Regimen
All-Cause Mortality (participants affected / at risk) | 11/223 | 8/112
Serious Adverse Events (participants affected / at risk) | 45/223 | 23/112
Other Adverse Events (participants affected / at risk) | 199/223 | 72/112
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | LAI + Multi-drug Regimen (N=223) | Multi-drug Regimen (N=112)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 6 (8) | 5 (7)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 7 (12) | 3 (3)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0)
Infective exacerbation of bronchiectasis (Infections and infestations) | 5 (8) | 3 (3)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1)
Cardiac failure (Cardiac disorders) | 1 (1) | 1 (1)
Cardiogenic shock (Cardiac disorders) | 0 (0) | 1 (1)
Microvascular coronary artery disease (Cardiac disorders) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (2) | 0 (0)
Pneumatosis intestinalis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Adenocarcinoma gastric (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Colon adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Breast cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Major depression (Psychiatric disorders) | 1 (1) | 0 (0)
Drug hypersensitivity (Immune system disorders) | 1 (1) | 1 (1)
Cachexia (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Spinal pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Peripheral vascular disorder (Vascular disorders) | 1 (1) | 0 (0)
Shock (Vascular disorders) | 1 (1) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Performance status decreased (General disorders) | 1 (1) | 0 (0)
Hepatic function abnormal (Hepatobiliary disorders) | 1 (1) | 0 (0)
Radius fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Computerised tomogram thorax abnormal (Investigations) | 1 (1) | 0 (0)
Urinary retention (Renal and urinary disorders) | 0 (0) | 1 (1)
Dermatitis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Anxiety (Psychiatric disorders) | 2 (2) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Pulmonary cavitation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0)
Alveolitis allergic (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Maxillary sinus pseudocyst (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Bronchial fistula (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Respiratory acidosis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 8 (9) | 2 (2)
Infective exacerbation of chronic obstructive airways disease (Infections and infestations) | 2 (2) | 1 (1)
Mycobacterium avium complex infection (Infections and infestations) | 1 (1) | 2 (2)
Lung infection (Infections and infestations) | 2 (4) | 0 (0)
Bronchitis (Infections and infestations) | 1 (1) | 0 (0)
Infectious pleural effusion (Infections and infestations) | 1 (1) | 0 (0)
Lung infection pseudomonal (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia pseudomonal (Infections and infestations) | 1 (1) | 0 (0)
Scedosporium infection (Infections and infestations) | 1 (1) | 0 (0)
Superinfection bacterial (Infections and infestations) | 1 (1) | 0 (0)
Mycetoma mycotic (Infections and infestations) | 0 (0) | 1 (1)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 2 (2)
Asthenia (General disorders) | 0 (0) | 1 (1)
Hypercapnic coma (Nervous system disorders) | 0 (0) | 1 (1)
Exostosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | LAI + Multi-drug Regimen (N=223) | Multi-drug Regimen (N=112)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 104 (140) | 2 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 85 (111) | 17 (20)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 47 (59) | 10 (10)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 37 (48) | 14 (17)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 24 (30) | 2 (2)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 15 (25) | 2 (3)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 15 (16) | 3 (4)
Infective exacerbation of bronchiectasis (Infections and infestations) | 15 (16) | 5 (6)
Nasopharyngitis (Infections and infestations) | 12 (15) | 8 (10)
Upper respiratory tract infection (Infections and infestations) | 8 (9) | 7 (10)
Diarrhoea (Gastrointestinal disorders) | 29 (31) | 5 (5)
Nausea (Gastrointestinal disorders) | 25 (30) | 4 (4)
Vomiting (Gastrointestinal disorders) | 14 (17) | 3 (4)
Constipation (Gastrointestinal disorders) | 6 (6) | 6 (6)
Fatigue (General disorders) | 36 (38) | 8 (8)
Pyrexia (General disorders) | 17 (22) | 5 (6)
Chest discomfort (General disorders) | 13 (13) | 3 (4)
Back pain (Musculoskeletal and connective tissue disorders) | 13 (15) | 4 (4)
Arthralgia (Musculoskeletal and connective tissue disorders) | 15 (16) | 3 (3)
Headache (Nervous system disorders) | 22 (25) | 5 (6)
Dizziness (Nervous system disorders) | 15 (16) | 3 (3)
Weight decreased (Investigations) | 18 (19) | 3 (3)
Tinnitus (Ear and labyrinth disorders) | 18 (22) | 1 (1)
Hypoacusis (Ear and labyrinth disorders) | 7 (7) | 6 (6)
Decreased appetite (Metabolism and nutrition disorders) | 15 (17) | 8 (8)
Pneumonia (Infections and infestations) | 2 (2) | 6 (6)
Sputum increased (Respiratory, thoracic and mediastinal disorders) | 13 (15) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Per the signed Investigator Agreement in the study protocol and protocol amendments, the PI agreed "not to originate or use the name of Insmed Incorporated, or study drug code in any publicity, news release, or other public announcement, written or oral, whether to the public, press, or otherwise, relating to this protocol, to any amendment to the protocol, or to the performance of this protocol, without the prior written consent of Insmed Incorporated."

DOCUMENTS (2):
  • Study Protocol (2016-02-22): https://cdn.clinicaltrials.gov/large-docs/04/NCT02344004/Prot_002.pdf
  • Statistical Analysis Plan (2016-10-24): https://cdn.clinicaltrials.gov/large-docs/04/NCT02344004/SAP_003.pdf